CLINICAL TRIAL: NCT05681078
Title: The Impact of Hearing Loss Severity on Balance Intervention Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 275305
Record Dates: First submitted 2022-12-21; First posted 2023-01-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2023-12

CONDITIONS: Hearing Loss; Fall; Postural Balance
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Matter of Balance Program (Experimental)
  Interventions: Behavioral: A Matter of Balance: Managing Concerns about Falls

INTERVENTIONS:
Behavioral: A Matter of Balance: Managing Concerns about Falls — A Matter of Balance is an evidence-based program targeting physical activity and fall prevention for adults 60 years of age and older. This program incorporates active learning discussions and activities along with exercise training to reduce the fear of falling, improve fall efficacy and management, and increase physical activity levels in older adults.

SUMMARY:
The goal of this study is to learn about how hearing loss impacts balance intervention outcomes and risk of falling in older adults. The main questions it aims to answer are:

* How does the evidence-based A Matter of Balance (AMOB) program affect older adults' falls risk and balance-related measures?
* Is the severity of someone's hearing loss related to their balance intervention (AMOB) outcomes?

Participants will:

* Complete a hearing and balance test
* Answer some questions about their background and health history, their thoughts about potential falls and how this impacts them, and their current physical activity level
* Participate in the A Matter of Balance Program, an evidence-based program that includes group discussion, activities, and exercises to reduce fall risk

ELIGIBILITY:
Inclusion Criteria:

* age of 60 years old or greater
* absence of any major physical or health condition that would prevent participation in the intervention sessions
* English speaking

Exclusion Criteria:

* severe balance disorder diagnosis
* uncorrected severe vision impairment

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in postural sway from baseline to after completion of AMOB | baseline and within 1 month post training
  Postural sway will be assessed using a Balance Tracking Systems pressure plate.

SECONDARY OUTCOMES:
Change in balance confidence from baseline to after completion of AMOB | baseline and within 1 month post training
  Assessed via the Activity-Specific Balance Confidence Scale. Each item is rated as a percentage reflecting an individual's level of confidence in being able to perform the activity without losing their balance (0% - no confidence, 100% - completely confident). The ratings are then averaged across the 16 items for the total score. A higher score suggests higher self confidence related to balance.
Change in falls risk from baseline to after completion of AMOB | baseline and within 1 month post training
  Assessed via Falls Risk Questionnaire. Point values are allocated to each questionnaire item (range: 0-14) with higher scores suggesting a greater falls risk.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT05681078/ICF_000.pdf